CLINICAL TRIAL: NCT02045186
Title: Monitoring of Oral HPV Infection in HPV-positive Oropharyngeal Squamous Cell Carcinoma During and After Chemoradiotherapy (CRT)
Brief Title: Monitoring of Oral Human Papillomavirus Infection (HPV) in HPV-positive Oropharyngeal Squamous Cell Carcinoma (OPSCC)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LCCC1338
Record Dates: First submitted 2014-01-22; First posted 2014-01-24 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Carcinoma, Squamous Cell; Head and Neck Neoplasms; Oropharyngeal Neoplasms
Keywords: Human Papilloma Virus; Oropharynx; Oropharyngeal Squamous Cell Carcinoma; Squamous Cell Carcinoma; Radiation Therapy; Chemotherapy
MeSH Terms: conditions — Carcinoma, Squamous Cell; Head and Neck Neoplasms; Oropharyngeal Neoplasms; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Assessment of Oral HPV Infection (Other): Oral HPV infection will be assessed 14 times, once prior to starting CRT, weekly during CRT, and then serially post-treatment: 4-8 weeks, 3 months, 6 months, 12 months, 18 months, 24 months. Patients will provide samples of their saliva and exfoliated epithelial cells at these timepoints. Samples will be collected with supplies provided by and analyzed by OralDNA Labs.
  Interventions: Other: Assessment of Oral HPV Infection

INTERVENTIONS:
Other: Assessment of Oral HPV Infection — Saliva and exfoliated oral epithelial cells will be collected with collection supplies provided by OralDNA Labs. Patients will swish and gargle a saline solution for 30 seconds and expectorate it into a funneled collection tube. The collected specimen will be sent to OralDNA Labs. Three diagnostic tests will be performed on each sample to assess oral HPV infection:
  1. Polymerase chain reaction (PCR) for HPV DNA.
  2. Fluorescent in-situ hybridization (FISH).
  3. Viral expression: The test is based on the measurement of the viral RNA levels by methods of detection of the fluorochrome labeled HPV probes by flow cytometry.

SUMMARY:
The purpose of this research study is to determine whether and when patients with human papilloma virus positive squamous cell cancer of the oropharynx treated with radiation and chemotherapy clear their human papilloma virus infection.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age (no upper age limit)
2. AnyT, AnyN, M0 squamous cell carcinoma of the oropharynx
3. Biopsy proven squamous cell carcinoma that is HPV positive via standard pathological assessment of tumor tissues in pathology department at the treating institution
4. Scheduled for definitive CRT as primary treatment of their oropharynx cancer

Exclusion Criteria:

1. Prior history of radiation therapy to the head and neck
2. Prior history of mucosal head and neck cancer.
3. Not willing or able to comply with study specific procedures

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-12; Primary Completion 2014-03 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with HPV-positive OPSCC undergoing CRT who are clear of their oral HPV infection at each time-point | 2 years post-CRT of last enrolled patient

SECONDARY OUTCOMES:
Time to HPV clearance for patients with HPV-positive OPSCC undergoing CRT | 2 years post-CRT of last enrolled patient
Number of aneuploidy cells as measured by FISH (Florescent in-situ hybridization) and the mRNA copy number for HPV E6 and HPV E7 at each time-point | 2 years post-CRT of last enrolled patient
Clinical outcomes of interest (local control, loco-regional control, distant metastasis-free survival, and overall survival (OS)) in patients with HPV-positive OPSCC undergoing CRT | 2 years post-CRT of last enrolled patient

CONTACTS AND LOCATIONS:
Overall Officials: Bhishamjit Chera, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Department of Radiation Oncology, Chapel Hill, North Carolina, United States